CLINICAL TRIAL: NCT04241458
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Oral Doses of BI 706321 in Healthy Male and Female Subjects (Doubleblind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Healthy Men and Women Tolerate Different Doses of BI 706321
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1425-0002; 2019-004351-36 (EudraCT Number)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 2 mg BI 706321 (Experimental): Subjects were orally administered a single daily dose of 2 x 1 capsule of 1 milligrams (mg) of BI 706321 on Day 1 and from Day 6 to 19. The trial medication was administered with about 240 millilitres (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 703621
- 5 mg BI 706321 (Experimental): Subjects were orally administered a single daily dose of 1 capsule of 5 milligrams (mg) of BI 706321 on Day 1 and from Day 6 to 19. The trial medication was administered with about 240 millilitres (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 703621
- 8 mg BI 706321 + 75 ug midazolam (Experimental): Subjects were orally administered a single daily dose of 1 capsule of 5 milligrams (mg) and 3 capsules of 1 mg of BI 706321 on Day 1 and from Day 6 to 19. Subjects were also orally administered a single daily dose of 1.5 millilitres (mL) (75 micrograms) of Midazolam solution on Day -1 and Day 19. The trial medication was administered with about 240 mL of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 703621; Drug: Midazolam
- 10 mg BI 706321+ 75 ug midazolam (Experimental): Subjects were orally administered a single daily dose of 2 capsules of 5 milligrams (mg) of BI 706321 on Day 1 and from Day 6 to 19. Subjects were also orally administered a single daily dose of 1.5 millilitres (mL) (75 micrograms) of Midazolam solution on Day -1 and Day 19. The trial medication was administered with about 240 mL of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 703621; Drug: Midazolam
- Placebo (Placebo Comparator): Subjects were orally administered a single daily dose of matching placebo to BI 706321 capsules on Day 1 and from Day 6 to 19. Three out of the seven subjects were also orally administered a single daily dose of 1.5 millilitres (mL) (75 micrograms) of Midazolam solution on Day -1 and Day 19. The trial medication was administered with about 240 millilitres (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 703621 — BI 703621
  Arms: 10 mg BI 706321+ 75 ug midazolam; 2 mg BI 706321; 5 mg BI 706321; 8 mg BI 706321 + 75 ug midazolam
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Midazolam — Midazolam
  Arms: 10 mg BI 706321+ 75 ug midazolam; 8 mg BI 706321 + 75 ug midazolam

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 706321 in healthy male and female subjects following oral administration of multiple rising doses for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), temperature), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive, at screening)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive, at screening)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR, temperature or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 45 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 30 days (or 5 half-lives (whichever longer)) of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker of more than 10 cigarettes or 3 cigars or 3 pipes per day
* Inability to refrain from smoking while in-house stay
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males), and unwillingness/inability to refrain from intake of alcoholic beverages from 48 hours prior to the trial medication administration and until Day 7 post trial medication administration.
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* ALT (alanine transaminase), AST (aspartate transaminase), or creatinine exceed upper limit of normal range at screening, confirmed by a repeat test
* hemoglobin (Hb), platelets and neutrophils below lower limit of normal range at screening, confirmed by a repeat test
* Positive result for human immunoinsufficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) infection at screening.
* History of tuberculosis (TB) or positive finding in interferon-gamma release assay (IGRA).

Female subjects will not be allowed to participate, if any of the following apply:

* Not surgically sterilised or not postmenopausal, defined as at least 1 year of spontaneous amenorrhea without an alternative medical cause (in questionable cases a blood sample with simultaneous levels of FSH above 30 U/L and estradiol below 20 ng/L is confirmatory)
* Positive pregnancy test
* Lactation

Male subjects will not be allowed to participate, if any of the following apply:

- Male subjects with women of childbearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of administration of trial medication until 30 days thereafter. Sperm donation is not allowed from the time point of drug administration until 30 days thereafter.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a double-blind, randomised, placebo-controlled, parallel group design trial in order to investigate safety, tolerability, and pharmacokinetics of BI 706321 in healthy male and female subjects following oral administration of multiple rising doses for 14 days.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
Started | 7 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received. The TS was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam | Total
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (8.7) | 49.1 (6.7) | 46.4 (8.9) | 42.5 (7.4) | 44.8 (7.6) | 44.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 1 | 0 | 4
  Male | 7 | 6 | 7 | 7 | 8 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 8 | 8 | 8 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 6 | 8 | 8 | 8 | 8 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events
Description: Number of subjects with drug-related adverse events is presented.
Time Frame: From first administration of study drug until 8 days after the last dosing, up to 27 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8
Participants | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 706321 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of BI 706321 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) is presented with a dosing interval τ of 24 hours. Pharmacokinetics parameters were determined after the last dose.
Time Frame: From 432.5 hours (h) and 433h, 434h, 435h, 436h, 437h, 438h, 440h, 442h, 444h, 446h, 456h after dosing on Day 1.
Population: Pharmacokinetic parameter analysis set (PKS):
  This set included all subjects in the treated set (TS) who provided at least 1 PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour(h)*nanomole(nmol)/Litre (L)
Arm/Group | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 7
hour(h)*nanomole(nmol)/Litre (L) | 88.1 (34.5) | 235 (34.8) | 517 (30.0) | 574 (35.6)

3. Secondary Outcome: Maximum Measured Concentration of BI 706321 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of BI 706321 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) is presented with a dosing interval τ of 24 hours. Pharmacokinetics parameters were determined after the last dose.
Time Frame: From 432.5 hours (h) and 433h, 434h, 435h, 436h, 437h, 438h, 440h, 442h, 444h, 446h and 456h after dosing on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole(nmol)/Litre(L)
Arm/Group | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 7
nanomole(nmol)/Litre(L) | 5.69 (41.8) | 14.7 (43.1) | 34.7 (38.5) | 39.9 (35.7)

4. Secondary Outcome: Minimum Concentration of BI 706321 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmin,ss)
Description: Minimum concentration of BI 706321 in plasma at steady state over a uniform dosing interval τ (Cmin,ss) is presented with a dosing interval τ of 24 hours. Pharmacokinetics parameters were determined after the last dose.
Time Frame: From 432.5 hours (h) and 433h, 434h, 435h, 436h, 437h, 438h, 440h, 442h, 444h, 446h and 456h after dosing on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole(nmol)/Litre(L)
Arm/Group | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 7
nanomole(nmol)/Litre(L) | 2.84 (31.0) | 7.29 (34.1) | 15.2 (28.3) | 17.3 (35.5)

5. Secondary Outcome: Accumulation Ratio Based on Cmax,ss (RA,Cmax)
Description: Accumulation ratio (RA) based on maximum measured concentration of BI 706321 in plasma at steady state over a uniform dosing interval τ (Cmax,ss), (RA,Cmax) is presented. RA,cmax = Cmax,ss [nmol/L]/ Cmax,1 [nmol/l], and the unit of measure is hence unitless.
Time Frame: Within 3 hours (h) prior to drug administration on Day 1 and 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h and 432.5h, 433h, 434h, 435h, 436h, 437h, 438h, 440h, 442h, 444h, 446h and 456h after dosing on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Unitless
Arm/Group | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 7
Unitless | 2.00 (27.7) | 2.28 (23.1) | 3.29 (24.5) | 3.34 (15.2)

6. Secondary Outcome: Accumulation Ratio Based on AUC0-τ (RA,AUC)
Description: Accumulation ratio (RA) based on area under the concentration-time curve of BI 706321 in plasma after repeated doses over the time interval from τ (AUC0-τ), (RA,AUC) is presented with a dosing interval τ of 24 hours.
  RA, AUC= AUC tau, ss [h*nmol/L]/ AUC tau,1 [h*nmol/L]; hence the unit of measure is unitless.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Untiless
Arm/Group | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 7
Untiless | 2.30 (33.3) | 2.76 (20.8) | 3.69 (23.9) | 3.58 (19.8)

ADVERSE EVENTS:
Time Frame: For on-treatment adverse events (AE) and all-cause mortality: From first administration of study drug until 8 days after the last dosing, up to 27 days.
Description: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received. The TS was used for safety analyses.
Arm/Group | Placebo | 2 mg BI 706321 | 5 mg BI 706321 | 8 mg BI 706321 + 75 ug Midazolam | 10 mg BI 706321+ 75 ug Midazolam
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/7 | 3/8 | 5/8 | 6/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | 2 mg BI 706321 (N=8) | 5 mg BI 706321 (N=8) | 8 mg BI 706321 + 75 ug Midazolam (N=8) | 10 mg BI 706321+ 75 ug Midazolam (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cheilosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 2 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT04241458/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT04241458/SAP_001.pdf